CLINICAL TRIAL: NCT02654288
Title: Dynamic Changes of the Serum Level of Immunoglobulin G4(IgG4) and Interleukin-10(IL-10) in the Patients of Pancreatic Cancer After Gemcitabine-based Chemotherapy
Brief Title: Dynamic Changes of Sera Immunoglobulin G4 and Interleukin-10 in the Patients of Pancreatic Cancer After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: 81272573
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Pancreatic Neoplasms; Inflammation
Keywords: pancreatic cancer; gemcitabine; chemotherapy; immunoglobulin G 4
MeSH Terms: conditions — Pancreatic Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The IgG4 in serum from peripheral blood will be detected.(4ml/test)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- single arm: The pancreatic cancer patients without history of chemotherapy who will receive gemcitabine-based chemotherapy will be recruited and the sera IgG4 and IL-10 will be detected before and after chemotherapy.
  Interventions: Other: gemcitabine-based chemotherapy

INTERVENTIONS:
Other: gemcitabine-based chemotherapy

SUMMARY:
Investigators have previously found that the infiltration of immunoglobulin G4(IgG4) positive plasma cells in tumor tissue predicts a poor prognosis of pancreatic cancer after curative resection. Investigators further attempt to explore the possible roles of IgG4 and the inducer of IgG4, interleukin-10(IL-10), in the chemotherapy of pancreatic cancer. In this primary study, investigators plan to observe the dynamic changes of sera IgG4 and IL-10 in peripheral blood after gemcitabine-based chemotherapy and analyze the correlations of IgG4 and IL-10 with the response of gemcitabine and overall survival of pancreatic cancer.

DETAILED DESCRIPTION:
Human immunoglobulin G(IgG) is a family consisting of four members, IgG1, IgG2, IgG3 and IgG4.IgG4 is regarded as an inhibitory IgG which can inhibit the activation of immune responses[1]. Recently it was reported that IgG4 could weaken the activation of macrophages to promote cancer progression[2]. Autoimmune pancreatitis(AIP) is the most common clinical manifestation of IgG4-related sclerosing diseases(IRSD) which is characterized by abundant infiltration of IgG4 positive plasma cells[3].Although there are abundant infiltrations of IgG4 positive plasma cells in pancreatic lesion of AIP, the correlation of IgG4 positive plasma cells with pancreatic cancer has never been reported.Investigators have previously found that higher level of infiltration of IgG4 positive plasma cells in tumor tissue predicts a poor prognosis of pancreatic cancer after curative resection(not published).Investigators further attempt to explore the possible roles of IgG4 and the inducer of IgG4, IL-10, in the chemotherapy of pancreatic cancer.Since gemcitabine is the first line chemotherapeutic drug for pancreatic cancer, in this primary study,investigators plan to observe the dynamic changes of sera IgG4 and IL-10 in peripheral blood after gemcitabine-based chemotherapy and analyze the correlations of IgG4 and IL-10 with the response of gemcitabine and overall survival of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 to 75-year old;
2. Pathological verified pancreatic cancer including adenocarcinoma and cancerogenesis of intraductal papillary mucinous neoplasm (IPMN);
3. Pancreatic cancer patients receiving adjuvant chemotherapy after curative resection; pancreatic cancer patients with recurrent lesions receiving chemotherapy after curative resection; pancreatic cancer patients with unresectable tumor receiving chemotherapy;
4. Patients have good physical status to receive chemotherapy;
5. No history of chemotherapy and the current regimen contains gemcitabine;
6. No medical history of IgG4 related diseases and other connective tissue diseases;
7. Written consent is available.

Exclusion Criteria:

1. Patient younger than 18-year old;
2. Patient has chemotherapy before;
3. The physical status is too poor to receive chemotherapy;
4. The patient has history of IgG4 related diseases and some other connective diseases;
5. Written consent is not available.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients without history of chemotherapy will be recruited. After evulation of the physical status, the patients will receive gemcitabine-based chemotherapy.The peripheral blood will be collected and the sera IgG4 and IL-10 will be detected during chemotherapy. Then the correlation of the dynamic changes of IgG4 and IL-10 with the response of chemotherapy and the overall survival will be analyzed.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The dynamic change patterns of sera IgG4 and IL-10 of pancreatic cancer after gemcitabine-based chemotherapy will be recorded. | one year
  Investigators attempt to analyze the dynamic change patterns of sera IgG4 and IL-10 of pancreatic cancer after gemcitabine-based chemotherapy and theoretically investigators imagine that the sera IgG4 and IL-10 will be elevated in most of the patients.

SECONDARY OUTCOMES:
The correlation of the changes of IgG4 and IL-10 with the tumor marker during chemotherapy will be analyzed | one year
  The sera IgG4 and IL-10 and tumor marker will be detected during chemotherapy and the correlations will be analyzed.
The correlation of the changes of IgG4 and IL-10 with the efficacy of chemotherapy evaluated by intravenous enhanced CT during chemotherapy will be analyzed | one year
  The sera IgG4 and IL-10 will be detected during chemotherapy and the chemotherapeutic efficacy will be evaluated by intravenous enhanced CT scan and the correlation will be analyzed.
The correlation of the changes of IgG4 and IL-10 with the overall survival after chemotherapy will be analyzed. | Two year
  The sera IgG4 and IL-10 will be detected during chemotherapy and the overall survival will be recorded and then the correlation will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Liao, MD, Principal Investigator — Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Davies AM, Sutton BJ. Human IgG4: a structural perspective. Immunol Rev. 2015 Nov;268(1):139-59. doi: 10.1111/imr.12349. PMID 26497518
- [Background] Karagiannis P, Villanova F, Josephs DH, Correa I, Van Hemelrijck M, Hobbs C, Saul L, Egbuniwe IU, Tosi I, Ilieva KM, Kent E, Calonje E, Harries M, Fentiman I, Taylor-Papadimitriou J, Burchell J, Spicer JF, Lacy KE, Nestle FO, Karagiannis SN. Elevated IgG4 in patient circulation is associated with the risk of disease progression in melanoma. Oncoimmunology. 2015 Jun 3;4(11):e1032492. doi: 10.1080/2162402X.2015.1032492. eCollection 2015 Nov. PMID 26451312
- [Background] Karagiannis P, Gilbert AE, Josephs DH, Ali N, Dodev T, Saul L, Correa I, Roberts L, Beddowes E, Koers A, Hobbs C, Ferreira S, Geh JL, Healy C, Harries M, Acland KM, Blower PJ, Mitchell T, Fear DJ, Spicer JF, Lacy KE, Nestle FO, Karagiannis SN. IgG4 subclass antibodies impair antitumor immunity in melanoma. J Clin Invest. 2013 Apr;123(4):1457-74. doi: 10.1172/JCI65579. PMID 23454746